CLINICAL TRIAL: NCT01647295
Title: Social Interactions: Ocular Explorations and Pupillometry in Autism
Acronym: ISEOP
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-60; 2012-A00520-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorders
Keywords: visual exploration; pupil size; social interactions; faces; human motion
MeSH Terms: conditions — Autism Spectrum Disorder; DiGeorge Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this work will first to characterize in typical childhood, visual exploratory behavior and pupillary response associated with salience of human social stimuli (faces and body movements), and then to evaluate these markers in children with autism.

The second objective of this work will be to achieve in a population of children with autism a longitudinal evaluation of these markers during development and therapeutics.

DETAILED DESCRIPTION:
Patients with autism have significant social difficulties and communication alterations. It has been shown in these patients difficulties to understand some clues indispensable to social relations, for example, faces and their emotions and motion of human bodies. The faces and human movements are an important source of information helping to interact with others. Understanding the intentions of the others through facial expressions and gestures can help them to adapt their behavior and their interactions. While in healthy subjects, faces and human movements receive special attention, autistic patients seem to pay less attention to this kind of social stimuli. It has already been shown that children and healthy adults spend more time looking at faces and human movements (relative to objects), whereas the opposite behavior is observed in patients with autism. Studying gaze behavior seems to be essential for progress in the understanding of autism pathology. Eye-tracking systems allow to measure precisely what a subject looks on a picture. Moreover, eye-tracking systems permit the measurement of the pupil size which variations are correlated with cognitive processes. The objective of this study is to analyze the ocular behavior (ocular scan path and pupil diameter) of young patients with autism when viewing faces and human movements and to compare these measurements with those of chronologically age-matched healthy children. This work will identify attentional problems concerning exploration of human faces and movements that can be related to their social difficulties. These disorders should be manifested by an atypical ocular scan path and by changes in pupil variation in response to face and human motion. Then to follow the evolution of these indices will allow to evaluate the effect of therapies. These results will highlight new data essential to understanding disorders of social relations and to better adapt rehabilitative strategies.

ELIGIBILITY:
Inclusion Criteria:

* For autistic children, diagnosis of autism spectrum disorders according to DSM IV-TR and ADI / ADOS criteria ; normal or corrected vision; no nervous system disease
* For healthy children, normal schooling and normal or corrected vision
* For all, parental consents

Exclusion Criteria:

* psychotropic treatment

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Autistic children from the University Hospital of Tours Healthy children from the normal population
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Total time spent on pictures | two years
  Total time tracked during exploration of faces and human motion, compared to objects

SECONDARY OUTCOMES:
Interest zones | two years
  Time spent on interest zones such as eyes or mouth.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Bretonneau, Tours, France

REFERENCES:
- [Result] Aguillon-Hernandez N, Mofid Y, Latinus M, Roche L, Bufo MR, Lemaire M, Malvy J, Martineau J, Wardak C, Bonnet-Brilhault F. The pupil: a window on social automatic processing in autism spectrum disorder children. J Child Psychol Psychiatry. 2020 Jul;61(7):768-778. doi: 10.1111/jcpp.13170. Epub 2019 Dec 11. PMID 31823380